CLINICAL TRIAL: NCT01595425
Title: A Phase I, Open-label, Randomized, Single-center, 2-way Crossover Bioequivalence Study Comparing a Pellets Based Sachet Formulation of D961H 20 mg and a Commercial HPMC Capsule of D961H 20 mg After Repeated Oral Administration in Japanese Healthy Male Subjects
Brief Title: Bioequivalence Study Comparing D961H Sachet and D961H Capsule in Japanese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D961TC00001
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Bioequivalence Study
Keywords: Bioequivalence,; pharmacokinetics,; safety,; esomeprazole,; Japanese,; healthy subject,; homo-EM
MeSH Terms: interventions — Esomeprazole

ARMS (2):
- D961H Sachet 20 mg (Experimental): 2 way crossover
  Interventions: Drug: D961H Sachet 20 mg
- D961HHPMC Capsule 20 mg (Experimental): 2 way crossover
  Interventions: Drug: D961H HPMC capsule 20 mg

INTERVENTIONS:
Drug: D961H Sachet 20 mg — Each volunteer will receive a D961H sachet 20 mg once in the morning for 5 days.
  Other Names: esomeprazole sachet
  Arms: D961H Sachet 20 mg
Drug: D961H HPMC capsule 20 mg — Each volunteer will receive a D961H HPMC capsule 20 mg once in the morning for 5 days.
  Other Names: esomeprazole; capsule 20 mg
  Arms: D961HHPMC Capsule 20 mg

SUMMARY:
This study is to investigate whether D961H sachet 20 mg is bioequivalent to D961H HPMC capsule 20 mg following repeated oral doses, and to evaluate the safety and tolerability of these two formulations in healthy male Japanese subjects.

DETAILED DESCRIPTION:
A Phase I, Open-label, Randomized, Single-center, 2-way Crossover Bioequivalence Study Comparing a Pellets Based Sachet Formulation of D961H 20 mg and a Commercial HPMC Capsule of D961H 20 mg After Repeated Oral Administration in Japanese Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures
2. Japanese healthy male subjects aged 20 to 45 years of age
3. Body Mass Index 19-27 kg/m2 and body weight 50-85 kg
4. Clinically normal findings
5. Classified as homo-EM(extensive metabolizers) according to the genotype of CYP2C19

Exclusion Criteria:

1. Significant clinical illness
2. Past or present cardiac, renal, hepatic, neurological or gastrointestinal disease
3. Clinical significant condition which could modify the absorption of the investigational product
4. Past or present severe allergic disease, hypersensitivity to food or drugs, or allergic symptoms requiring medical intervention

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
AUCτ and Cmax,ss of D961H | Day 5
  * AUC(0-t)-Area under plasma concentration time curve from zero to time of the last measurable concentration
  * Cmax,ss - maximum concentration at steady state

SECONDARY OUTCOMES:
Profile of pharmacokinetic of D961H in terms of AUC0-t,ss, MRT, tmax,ss, and t1/2. | Day 5
  * AUC0-t,ss-Area under plasma concentration time curve from zero to time of the last measurable concentration at steady state
  * MRT- Mean residence time
  * tmax,ss -time of maximum concentration at steady state
  * t½ -Terminal half-life
Safety and tolerability of a D961H in terms of clinical laboratory tests, blood pressure, pulse rate and body temperature. | Up to 5 to 7 days after the last dose.
Number of participants with adverse events. | Up to 5 to 7 days after the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Masataka Date, Study Director — AstraZeneca R&D Japan; Masanari Shiramoto, Principal Investigator — Hakata Clinic
Locations (1):
- Research Unit, Fukuoka, Fukuoka, Japan